CLINICAL TRIAL: NCT01148225
Title: A Multicenter Open-Label Study of the Long-term Safety and Efficacy of the Human Anti-TNF Monoclonal Antibody Adalimumab in Subjects With Non-infectious Intermediate Uveitis, Posterior Uveitis, or Panuveitis
Brief Title: A Study of the Long-term Safety and Efficacy of Adalimumab in Subjects With Intermediate-, Posterior-, or Pan-uveitis
Acronym: VISUAL III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M11-327; 2009-016196-29 (EudraCT Number)
Record Dates: First submitted 2010-05-14; First posted 2010-06-22 (Estimated); Results first posted 2019-04-04 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Uveitis
Keywords: Intermediate-Uveitis; Non-infectious Uveitis; Posterior-Uveitis; Active Uveitis; Pan-uveitis; Uveitis
MeSH Terms: conditions — Uveitis; Uveitis, Intermediate; Uveitis, Posterior | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Adalimumab (Other): Participants received open label (OL) adalimumab 40 mg by subcutaneous (SC) injection every other week (eow) until the final visit.
  Interventions: Drug: adalimumab

INTERVENTIONS:
Drug: adalimumab — Adalimumab, pre-filled syringe, administered by SC injection
  Other Names: ABT-D2E7; Humira

SUMMARY:
The purpose of this study is to evaluate the long term efficacy and safety of adalimumab participants with non-infectious intermediate-, posterior- or pan-uveitis.

DETAILED DESCRIPTION:
This study was initially planned to run for 78 weeks but was extended for ethical reasons, to avoid leaving participants untreated who had responded well to adalimumab treatment, so that participants were allowed to remain in the study until regulatory and/or reimbursement approval for the treatment of uveitis in adults was obtained for their respective countries. Data were collected through Week 366 (maximum), but because of decreasing sample size that became too small toward the end of the study to allow for meaningful conclusion, data cut off for efficacy analyses (intent to treat [ITT] population) occurred at Week 246, as less than 10% of participants in the ITT set had visits beyond this timepoint.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have successfully enrolled in either study M10-877 or M10-880 and either met the endpoint of "Treatment Failure" or completed the study

Exclusion Criteria:

* A participant will be excluded from this study if the participant discontinued from study M10-877 or M10-880 for any reasons other than having a Treatment Failure event
* Participant with corneal or lens opacity that precludes visualization of the fundus or that likely requires cataract surgery during the duration of the trial
* Participants with intraocular pressure of >= 25 mmHg and on >= 2 glaucoma medications or evidence of glaucomatous optic nerve injury
* Participant with proliferative or severe non-proliferative diabetic retinopathy or clinically significant macular edema due to diabetic retinopathy
* Participant with neovascular/wet age-related macular degeneration
* Participant with abnormality of vitreo-retinal interface (i.e., vitreomacular traction, epiretinal membranes, etc.) with the potential for macular structural damage independent of the inflammatory process
* Participant with a systemic inflammatory disease that requires therapy with a prohibited immunosuppressive agent at the time of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2010-11-23 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Suhler EB, Jaffe GJ, Fortin E, Lim LL, Merrill PT, Dick AD, Brezin AP, Nguyen QD, Thorne JE, Van Calster J, Cimino L, Adan A, Goto H, Kaburaki T, Kramer M, Vitale AT, Kron M, Song AP, Liu J, Pathai S, Douglas KM, Schlaen A, Muccioli C, Van Velthoven MEJ, Zierhut M, Rosenbaum JT. Long-Term Safety and Efficacy of Adalimumab in Patients with Noninfectious Intermediate Uveitis, Posterior Uveitis, or Panuveitis. Ophthalmology. 2021 Jun;128(6):899-909. doi: 10.1016/j.ophtha.2020.10.036. Epub 2020 Nov 3. PMID 33157077
- See also: This clinical study may be evaluating a usage that is not currently FDA-approved. Please see US Prescribing Information for approved uses. — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 424 participants were enrolled and received ≥1 dose of study drug (Safety population); 364 participants were included in the intent-to-treat (ITT) population (reasons for exclusion: incomplete efficacy data or GCP compliance issues at 2 sites (n=7); diabetic retinopathy [n=1]; cataract surgery [n=26]; and previous vitrectomy [n=26]).
Period: Overall Study
Arm/Group | Adalimumab
Started | 424
Completed | 239
Not Completed | 185
Not completed — Other | 185

BASELINE CHARACTERISTICS:
Population: Safety population
Arm/Group | Adalimumab
Number analyzed (Participants) | 424
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.44 (14.066)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 249
  Male | 175
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 77
  Not Hispanic or Latino | 347
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent events (TEAEs/TESAEs) are defined as any event with an onset date on or after the first dose of study drug and up to 70 days after the last dose. See the Adverse Event section for details.
Time Frame: Baseline to Final Visit (up to 366 weeks)
Population: Safety analysis set: includes all participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 424
participants
  Any TEAE | 398
  Any TESAE | 101

2. Primary Outcome: Hematology: Number of Participants With Potentially Clinically Significant (PCS) Values
Description: PCS laboratory values were defined as Common Toxicity Criteria (CTC) according to the National Cancer Institute Common Terminology for Adverse Events (NCI CTCAE) v3.0 ≥ Grade 3. Abbreviations used include g=grams; L=liters.
Time Frame: Baseline to Final Visit (Up to 366 weeks)
Population: Safety analysis set.
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 424
participants
  Hemoglobin (Low: <80-65 g/L) | 3
  Neutrophils (Low: <1.0-0.5*10^9/L) | 6
  Lymphocytes (Low: <0.5-0.2*10^9/L) | 7

3. Primary Outcome: Chemistry: Number of Participants With PCS Values
Description: PCS laboratory values were defined as Common Toxicity Criteria (CTC) according to the National Cancer Institute Common Terminology for Adverse Events (NCI CTCAE) v3.0 ≥ Grade 3. Abbreviations include ALT/SGPT=alanine aminotransferase/serum glutamate pyruvate transaminase; AST/SGOT=aspartate aminotransferase/serum glutamate oxaloacetate transaminase; g/L=grams/liter; mmol/L=millimoles/liter; ULN=upper limit of normal.
Time Frame: Baseline to Final Visit (Up to 366 weeks)
Population: Safety analysis set.
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 424
participants
  ALT/SGPT (High: >5.0-20.0*ULN) | 2
  AST/SGOT (High: >5.0-20.0*ULN) | 3
  Bilirubin, Total (High: >3.0-10.0*ULN) | 1
  Creatinine (High: >3.0-6.0*ULN) | 2
  Phosphate Inorganic (Low:<0.6-0.3 mmol/L) | 5
  Sodium (Low: <130-120 mmol/L) | 4
  Potassium (Low:<3.0-2.5 mmol/L) | 7
  Glucose (High: >13.9-27.8 mmol/L) | 18
  Albumin (Low: <20.0 g/L) | 2
  Cholesterol (High: >10.34-12.92 mmol/L) | 3
  Triglycerides (High: >5.0-10*ULN) | 8

4. Primary Outcome: Pulse (Sitting): Mean Change (Beats Per Minute) From Baseline To Final Visit
Description: Heart rate (beats per minute) was measured while the participant was sitting.
Time Frame: Baseline to Final Visit (Up to 366 weeks)
Population: Safety analysis set.
Measure: Mean (Standard Deviation); unit: beats per minute
Groups:
- Adalimumab: Participants received open label (OL) adalimumab 40 mg by subcutaneous injection(SC) every other week (eow) until the final visit.
Arm/Group | Adalimumab
Number analyzed (Participants) | 424
beats per minute | -1.0 (11.92)

5. Primary Outcome: Respiratory Rate (Sitting): Mean Change (Respirations Per Minute) From Baseline To Final Visit
Description: Respiratory rate (respirations per minute) was measured while the participant was sitting.
Time Frame: Baseline to Final Visit (Up to 366 weeks)
Population: Safety analysis set.
Measure: Mean (Standard Deviation); unit: respirations per minute
Arm/Group | Adalimumab
Number analyzed (Participants) | 424
respirations per minute | -0.1 (2.94)

6. Primary Outcome: Temperature (Sitting): Mean Change (Centigrade) From Baseline To Final Visit
Description: Temperature was measured while the participant was sitting.
Time Frame: Baseline to Final Visit (Up to 366 weeks)
Population: Safety analysis set.
Measure: Mean (Standard Deviation); unit: Centigrade
Arm/Group | Adalimumab
Number analyzed (Participants) | 424
Centigrade | -0.03 (0.516)

7. Primary Outcome: Diastolic and Systolic Blood Pressure (Sitting): Mean Change (mmHg) From Baseline To Final Visit
Description: Blood pressure was measured while the participant was sitting. Abbreviations used include mmHg=millimeters of mercury.
Time Frame: Baseline to Final Visit (Up to 366 weeks)
Population: Safety analysis set.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Adalimumab
Number analyzed (Participants) | 424
mmHg
  Diastolic Blood Pressure (Sitting) | 1.443 (10.4373)
  Systolic Blood Pressure (Sitting) | 1.955 (14.6281)

8. Secondary Outcome: Percentage of Participants in Quiescence Over Time
Description: Quiescence is defined as no active inflammatory lesions and anterior chamber (AC) cell grade ≤ 0.5+ and vitreous haze (VH) grade ≤0.5+. Participants with active uveitis at study entry could have been in quiescence at Week 0 because all participants were evaluated for uveitis status at the Final/Early Termination visit of the lead-in study and the Week 0 visit could have occurred up to 28 days later during which time the participant's disease status may have changed.
Time Frame: Weeks 0, 2, 4, 8, 12, 18, 30, 42, 54, 66, 78, 90, 102, 114, 126, 138, 150, 162, 174, 186, 198, 210, 222, 234, and 246
Population: ITT analysis set: includes all participants who received at least one dose of study medication with evaluable data at a given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Adalimumab: Participants received open label (OL) adalimumab 40 mg by subcutaneous injection (SC) every other week (eow) until the final visit.
Arm/Group | Adalimumab
Number analyzed (Participants) | 364
percentage of participants
  Week 0 | 33.5 [28.7 to 38.6]
  Week 2: number analyzed (Participants) | 348
  Week 2 | 56.3 [50.9 to 61.6]
  Week 4: number analyzed (Participants) | 323
  Week 4 | 63.8 [58.3 to 69.0]
  Week 8: number analyzed (Participants) | 343
  Week 8 | 72.0 [66.9 to 76.7]
  Week 12: number analyzed (Participants) | 333
  Week 12 | 72.4 [67.2 to 77.1]
  Week 18: number analyzed (Participants) | 330
  Week 18 | 75.2 [70.1 to 79.7]
  Week 30: number analyzed (Participants) | 319
  Week 30 | 79.9 [75.1 to 84.2]
  Week 42: number analyzed (Participants) | 310
  Week 42 | 81.3 [76.5 to 85.5]
  Week 54: number analyzed (Participants) | 296
  Week 54 | 81.1 [76.1 to 85.4]
  Week 66: number analyzed (Participants) | 284
  Week 66 | 85.9 [81.3 to 89.7]
  Week 78: number analyzed (Participants) | 271
  Week 78 | 86.3 [81.7 to 90.2]
  Week 90: number analyzed (Participants) | 261
  Week 90 | 87.4 [82.7 to 91.1]
  Week 102: number analyzed (Participants) | 245
  Week 102 | 87.3 [82.5 to 91.2]
  Week 114: number analyzed (Participants) | 231
  Week 114 | 87.9 [83.0 to 91.8]
  Week 126: number analyzed (Participants) | 215
  Week 126 | 88.4 [83.3 to 92.3]
  Week 138: number analyzed (Participants) | 196
  Week 138 | 89.3 [84.1 to 93.2]
  Week 150: number analyzed (Participants) | 180
  Week 150 | 85.0 [78.9 to 89.9]
  Week 162: number analyzed (Participants) | 154
  Week 162 | 87.0 [80.7 to 91.9]
  Week 174: number analyzed (Participants) | 142
  Week 174 | 87.3 [80.7 to 92.3]
  Week 186: number analyzed (Participants) | 128
  Week 186 | 90.6 [84.2 to 95.1]
  Week 198: number analyzed (Participants) | 113
  Week 198 | 89.4 [82.2 to 94.4]
  Week 210: number analyzed (Participants) | 88
  Week 210 | 88.6 [80.1 to 94.4]
  Week 222: number analyzed (Participants) | 70
  Week 222 | 92.9 [84.1 to 97.6]
  Week 234: number analyzed (Participants) | 51
  Week 234 | 96.1 [86.5 to 99.5]
  Week 246: number analyzed (Participants) | 42
  Week 246 | 95.2 [83.8 to 99.4]

9. Secondary Outcome: Percentage of Participants With Uveitis Flare Among Participants With Inactive Uveitis at Study Start
Description: Uveitis flare is defined as no quiescence (active inflammatory lesions and AC cell grade > 0.5+ and/or VH grade >0.5+).
Time Frame: 366 Weeks
Population: All participants in the ITT analysis set with inactive uveitis with evaluable data at a given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 124
percentage of participants | 38.7 [30.1 to 47.9]

10. Secondary Outcome: Percentage of Participants With Uveitis Flare From Week 8 Through Last Visit Among Participants With Active Uveitis at Study Start
Description: Uveitis flare is defined as no quiescence (active inflammatory lesions and AC cell grade > 0.5+ and/or VH grade >0.5+).
Time Frame: Weeks 8 to 246 (238 Weeks)
Population: All participants in the ITT analysis set with active uveitis at study start with evaluable data at a given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 232
percentage of participants | 67.7 [61.2 to 73.6]

11. Secondary Outcome: Percentage of Participants With New Active Inflammatory Lesions or Grade ≥2 in Anterior Chamber (AC) Cells or Grade ≥2 in Vitreous Haze (VH) Over Time
Description: Dilated indirect ophthalmoscopy is performed to determine both vitreous haze grading and the absence/presence of inflammatory chorioretinal and/or inflammatory retinal vascular lesions. The number of AC cells observed within a 1 mm * 1 mm slit beam was recorded for each eye and this number was used to determine the grade according to Standardization of Uveitis Nomenclature (SUN) criteria. Grading of VH was based on the National Eye Institute (NEI) publication which was adapted by the SUN working group. The percentage of participants with new active inflammatory lesions or grade ≥2 in AC cells or grade ≥2 in VH are presented.
Time Frame: Weeks 2, 4, 8, 12, 18, 30, 42, 54, 66, 78, 90, 102, 114, 126, 138, 150, 162, 174, 186, 198, 210, 222, 234, and 246
Population: All participants in the ITT analysis set with evaluable data at a given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 364
percentage of participants
  Week 2: number analyzed (Participants) | 348
  Week 2 | 11.8 [8.6 to 15.6]
  Week 4: number analyzed (Participants) | 323
  Week 4 | 8.4 [5.6 to 11.9]
  Week 8: number analyzed (Participants) | 343
  Week 8 | 7.6 [5.0 to 10.9]
  Week 12: number analyzed (Participants) | 333
  Week 12 | 6.9 [4.4 to 10.2]
  Week 18: number analyzed (Participants) | 330
  Week 18 | 3.6 [1.9 to 6.3]
  Week 30: number analyzed (Participants) | 319
  Week 30 | 5.3 [3.1 to 8.4]
  Week 42: number analyzed (Participants) | 310
  Week 42 | 4.2 [2.3 to 7.1]
  Week 54: number analyzed (Participants) | 296
  Week 54 | 4.1 [2.1 to 7.0]
  Week 66: number analyzed (Participants) | 284
  Week 66 | 1.4 [0.4 to 3.6]
  Week 78: number analyzed (Participants) | 271
  Week 78 | 4.1 [2.0 to 7.1]
  Week 90: number analyzed (Participants) | 261
  Week 90 | 4.6 [2.4 to 7.9]
  Week 102: number analyzed (Participants) | 245
  Week 102 | 4.1 [2.0 to 7.4]
  Week 114: number analyzed (Participants) | 231
  Week 114 | 4.8 [2.4 to 8.4]
  Week 126: number analyzed (Participants) | 215
  Week 126 | 3.3 [1.3 to 6.6]
  Week 138: number analyzed (Participants) | 196
  Week 138 | 2.0 [0.6 to 5.1]
  Week 150: number analyzed (Participants) | 180
  Week 150 | 4.4 [1.9 to 8.6]
  Week 162: number analyzed (Participants) | 154
  Week 162 | 3.2 [1.1 to 7.4]
  Week 174: number analyzed (Participants) | 142
  Week 174 | 1.4 [0.2 to 5.0]
  Week 186: number analyzed (Participants) | 128
  Week 186 | 1.6 [0.2 to 5.5]
  Week 198: number analyzed (Participants) | 113
  Week 198 | 0 [0 to 0]
  Week 210: number analyzed (Participants) | 88
  Week 210 | 3.4 [0.7 to 9.6]
  Week 222: number analyzed (Participants) | 70
  Week 222 | 1.4 [0 to 7.7]
  Week 234: number analyzed (Participants) | 51
  Week 234 | 0 [0 to 0]
  Week 246: number analyzed (Participants) | 42
  Week 246 | 0 [0 to 0]

12. Secondary Outcome: Percentage of Participants With Steroid-free Quiescence Over Time
Description: Steroid-free quiescence is defined as no active inflammatory lesions and AC cell grade ≤ 0.5+ and VH grade ≤0.5+ and no uveitis-related corticosteroids on the day of assessment.
Time Frame: Weeks 0, 2, 4, 8, 12, 18, 30, 42, 54, 66, 78, 90, 102, 114, 126, 138, 150, 162, 174, 186, 198, 210, 222, 234, and 246
Population: All participants in the ITT analysis set in steroid-free quiescence with evaluable data at a given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 364
percentage of participants
  Week 0 | 30.5 [25.8 to 35.5]
  Week 2: number analyzed (Participants) | 348
  Week 2 | 34.8 [29.8 to 40.0]
  Week 4: number analyzed (Participants) | 323
  Week 4 | 35.6 [30.4 to 41.1]
  Week 8: number analyzed (Participants) | 343
  Week 8 | 41.4 [36.1 to 46.8]
  Week 12: number analyzed (Participants) | 333
  Week 12 | 44.4 [39.0 to 50.0]
  Week 18: number analyzed (Participants) | 330
  Week 18 | 47.6 [42.1 to 53.1]
  Week 30: number analyzed (Participants) | 319
  Week 30 | 52.4 [46.7 to 57.9]
  Week 42: number analyzed (Participants) | 310
  Week 42 | 55.8 [50.1 to 61.4]
  Week 54: number analyzed (Participants) | 296
  Week 54 | 55.7 [49.9 to 61.5]
  Week 66: number analyzed (Participants) | 284
  Week 66 | 56.7 [50.7 to 62.5]
  Week 78: number analyzed (Participants) | 272
  Week 78 | 57.7 [51.6 to 63.7]
  Week 90: number analyzed (Participants) | 261
  Week 90 | 60.2 [53.9 to 66.1]
  Week 102: number analyzed (Participants) | 245
  Week 102 | 65.7 [59.4 to 71.6]
  Week 114: number analyzed (Participants) | 231
  Week 114 | 66.2 [59.7 to 72.3]
  Week 126: number analyzed (Participants) | 215
  Week 126 | 66.0 [59.3 to 72.3]
  Week 138: number analyzed (Participants) | 196
  Week 138 | 67.9 [60.8 to 74.3]
  Week 150: number analyzed (Participants) | 180
  Week 150 | 65.0 [57.6 to 71.9]
  Week 162: number analyzed (Participants) | 154
  Week 162 | 63.0 [54.8 to 70.6]
  Week 174: number analyzed (Participants) | 142
  Week 174 | 65.5 [57.1 to 73.3]
  Week 186: number analyzed (Participants) | 128
  Week 186 | 68.0 [59.1 to 75.9]
  Week 198: number analyzed (Participants) | 113
  Week 198 | 64.6 [55.0 to 73.4]
  Week 210: number analyzed (Participants) | 89
  Week 210 | 64.0 [53.2 to 73.9]
  Week 222: number analyzed (Participants) | 71
  Week 222 | 69.0 [56.9 to 79.5]
  Week 234: number analyzed (Participants) | 51
  Week 234 | 78.4 [64.7 to 88.7]
  Week 246: number analyzed (Participants) | 42
  Week 246 | 83.3 [68.6 to 93.0]

13. Secondary Outcome: Percentage of Participants in Non-quiescence (With/Without Change in Concomitant Medications Within 5 Days and With/Without Quiescence at Next Visit at Least 8 Weeks After Non-quiescence) Among Participants With Inactive Uveitis at Study Start
Description: Percentage of participants, without quiescence, with/without change in concomitant medications within 5 days after non-quiescence and with/without quiescence at next visit at least 8 weeks after non-quiescence among participants with inactive uveitis at study start. Quiescence is defined as no active inflammatory lesions and AC cell grade ≤ 0.5+ and VH grade ≤0.5+. Abbreviations used are as follows: CM=concomitant medications; NQ=non-quiescence.
Time Frame: 366 Weeks
Population: All participants in the ITT analysis set with inactive uveitis at Week 0 in nonquiescence with evaluable data at a given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 124
percentage of participants
  NQ With CM Change and quiescence at next visit | 10.5
  NQ With CM Change and nonquiescence at next visit | 2.4
  NQ Without CM Change and quiescence at next visit | 13.7
  NQ Without CM Change and NQ at next visit | 8.9
  NQ With Premature Discontinuation | 3.2
  NQ And Completion | 0.8

14. Secondary Outcome: Percentage of Participants in Non-quiescence (With/Without Change in Concomitant Medications Within 5 Days and With/Without Quiescence at Next Visit at Least 8 Weeks After Non-quiescence) Among Participants With Active Uveitis at Study Start
Description: Percentage of participants, without quiescence, with/without change in concomitant medications within 5 days after non-quiescence and with/without quiescence at next visit at least 8 weeks after non-quiescence, among participants with active uveitis at study start. Quiescence is defined as no active inflammatory lesions and AC cell grade ≤ 0.5+ and VH grade ≤0.5+. Abbreviations used include: CM=concomitant medications, NQ=non-quiescence.
Time Frame: 366 Weeks
Population: All participants in the ITT analysis set with active uveitis at Week 0 in nonquiescence with evaluable data at a given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 240
percentage of participants
  NQ With CM Change and quiescence at next visit | 19.2
  NQ With CM Change and nonquiescence at next visit | 10.8
  NQ Without CM Change and quiescence at next visit | 15.0
  NQ Without CM Change and NQ at next visit | 15.4
  NQ With Premature Discontinuation | 6.7
  NQ And Completion | 0.4

15. Secondary Outcome: Percentage of Participants Who Started Uveitis-related Systemic Corticosteroids During the Study
Description: Percentage of participants who started uveitis-related systemic corticosteroids during the study.
Time Frame: 366 Weeks
Population: All participants in the ITT analysis set without systemic corticosteroids at baseline with evaluable data at a given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 364
percentage of participants | 20.3 [16.3 to 24.8]

16. Secondary Outcome: Mean Daily Dose in Milligrams (mg) of Uveitis-related Systemic Corticosteroids in Participants With Active Uveitis Over Time
Description: Corticosteroid doses were converted into prednisone equivalents. Participants with uveitis-related systemic corticosteroid that could not be converted to prednisone equivalents were excluded. Individual mean daily doses were calculated within the respective visit windows. For Week 0, only uveitis-related systemic corticosteroids at Baseline (Day 1 for all participants) were considered. Baseline was defined as Week 0 for all participants.
Time Frame: Weeks 0, 2, 4, 8, 12, 18, 30, 42, 54, 66, 78, 90, 102, 114, 126, 138, 150, 162, 174, 186, 198, 210, 222, 234, and 246
Population: All participants in the ITT analysis set with active uveitis with a daily dose of uveitis-related systemic corticosteroids with evaluable data at a given timepoint.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Adalimumab
Number analyzed (Participants) | 235
milligrams
  Week 0 | 13.6 (19.21)
  Week 2 | 14.8 (17.12)
  Week 4: number analyzed (Participants) | 230
  Week 4 | 10.1 (12.27)
  Week 8: number analyzed (Participants) | 227
  Week 8 | 7.3 (9.75)
  Week 12: number analyzed (Participants) | 222
  Week 12 | 6.0 (9.34)
  Week 18: number analyzed (Participants) | 216
  Week 18 | 5.1 (8.47)
  Week 30: number analyzed (Participants) | 207
  Week 30 | 4.4 (7.12)
  Week 42: number analyzed (Participants) | 196
  Week 42 | 3.5 (5.54)
  Week 54: number analyzed (Participants) | 188
  Week 54 | 3.5 (6.71)
  Week 66: number analyzed (Participants) | 179
  Week 66 | 3.1 (6.32)
  Week 78: number analyzed (Participants) | 171
  Week 78 | 2.6 (5.10)
  Week 90: number analyzed (Participants) | 164
  Week 90 | 2.2 (4.47)
  Week 102: number analyzed (Participants) | 155
  Week 102 | 2.1 (4.80)
  Week 114: number analyzed (Participants) | 148
  Week 114 | 1.8 (4.50)
  Week 126: number analyzed (Participants) | 139
  Week 126 | 1.6 (4.16)
  Week 138: number analyzed (Participants) | 132
  Week 138 | 2.2 (5.65)
  Week 150: number analyzed (Participants) | 122
  Week 150 | 2.0 (4.49)
  Week 162: number analyzed (Participants) | 115
  Week 162 | 1.9 (4.31)
  Week 174: number analyzed (Participants) | 109
  Week 174 | 1.9 (4.46)
  Week 186: number analyzed (Participants) | 96
  Week 186 | 1.6 (4.27)
  Week 198: number analyzed (Participants) | 86
  Week 198 | 1.6 (4.05)
  Week 210: number analyzed (Participants) | 74
  Week 210 | 1.4 (3.57)
  Week 222: number analyzed (Participants) | 59
  Week 222 | 2.3 (8.48)
  Week 234: number analyzed (Participants) | 42
  Week 234 | 1.1 (3.17)
  Week 246: number analyzed (Participants) | 35
  Week 246 | 0.6 (1.69)

17. Secondary Outcome: Mean Daily Dose (mg) of Uveitis-related Systemic Corticosteroids in Participants With Inactive Uveitis Over Time
Description: as for outcome 16
Time Frame: Weeks 0, 2, 4, 8, 12, 18, 30, 42, 54, 66, 78, 90, 102, 114, 126, 138, 150, 162, 174, 186, 198, 210, 222, 234, and 246
Population: All participants in the ITT analysis set with inactive uveitis with a daily dose of uveitis-related systemic corticosteroids with evaluable data at a given timepoint.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Adalimumab
Number analyzed (Participants) | 124
milligrams
  Week 0 | 1.5 (7.32)
  Week 2 | 1.6 (6.65)
  Week 4: number analyzed (Participants) | 123
  Week 4 | 1.4 (4.89)
  Week 8: number analyzed (Participants) | 117
  Week 8 | 0.9 (3.41)
  Week 12: number analyzed (Participants) | 115
  Week 12 | 0.9 (4.12)
  Week 18: number analyzed (Participants) | 114
  Week 18 | 0.8 (3.29)
  Week 30: number analyzed (Participants) | 113
  Week 30 | 0.7 (2.74)
  Week 42: number analyzed (Participants) | 112
  Week 42 | 0.7 (2.64)
  Week 54: number analyzed (Participants) | 108
  Week 54 | 1.8 (7.09)
  Week 66: number analyzed (Participants) | 103
  Week 66 | 1.3 (5.32)
  Week 78: number analyzed (Participants) | 99
  Week 78 | 1.1 (4.36)
  Week 90: number analyzed (Participants) | 95
  Week 90 | 1.2 (4.54)
  Week 102: number analyzed (Participants) | 91
  Week 102 | 0.6 (2.63)
  Week 114: number analyzed (Participants) | 84
  Week 114 | 0.6 (2.67)
  Week 126: number analyzed (Participants) | 77
  Week 126 | 0.7 (2.95)
  Week 138: number analyzed (Participants) | 64
  Week 138 | 0.5 (2.09)
  Week 150: number analyzed (Participants) | 59
  Week 150 | 0.5 (1.91)
  Week 162: number analyzed (Participants) | 39
  Week 162 | 0.2 (1.00)
  Week 174: number analyzed (Participants) | 34
  Week 174 | 0.2 (1.07)
  Week 186: number analyzed (Participants) | 31
  Week 186 | 0.3 (1.12)
  Week 198: number analyzed (Participants) | 26
  Week 198 | 0.3 (1.23)
  Week 210: number analyzed (Participants) | 16
  Week 210 | 0.4 (1.50)
  Week 222: number analyzed (Participants) | 12
  Week 222 | 0.5 (1.73)
  Week 234: number analyzed (Participants) | 9
  Week 234 | 0.5 (1.57)
  Week 246: number analyzed (Participants) | 7
  Week 246 | 0.0 (0.00)

18. Secondary Outcome: Percent Change in Mean Daily Dose of Uveitis-related Systemic Corticosteroids Relative to Week 0 in Participants With Inactive Uveitis Using Systemic Corticosteroids at Week 0 Over Time
Description: Corticosteroid doses were converted into prednisone equivalents. Participants with uveitis-related systemic corticosteroid that could not be converted to prednisone equivalents were excluded. Individual mean daily doses were calculated within the respective visit windows. For Week 0, only uveitis-related systemic corticosteroids at Baseline (Day 1 for all participants) were considered. Baseline was defined as Week 0 for all participants. Data not presented after Week 198 as no participants remained on study as of Week 198.
Time Frame: Weeks 0, 2, 4, 8, 12, 18, 30, 42, 54, 66, 78, 90, 102, 114, 126, 138, 150, 162, 174, 186, and 198
Population: All participants in the ITT analysis set who received systemic corticosteroids at Week 0 with evaluable data at a given timepoint.
Measure: Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Adalimumab
Number analyzed (Participants) | 7
percent change from baseline
  Week 2 | -11.8 [-21.6 to -2.1]
  Week 4 | -46.6 [-64.2 to -29.0]
  Week 8 | -64.5 [-88.1 to -40.8]
  Week 12 | -29.7 [-91.5 to 32.1]
  Week 18 | -30.8 [-128.4 to 66.7]
  Week 30: number analyzed (Participants) | 6
  Week 30 | -25.0 [-159.6 to 109.5]
  Week 42: number analyzed (Participants) | 6
  Week 42 | -36.7 [-150.4 to 76.9]
  Week 54: number analyzed (Participants) | 5
  Week 54 | -11.9 [-186.2 to 162.5]
  Week 66: number analyzed (Participants) | 5
  Week 66 | -25.1 [-156.9 to 106.6]
  Week 78: number analyzed (Participants) | 5
  Week 78 | -28.3 [-157.9 to 101.2]
  Week 90: number analyzed (Participants) | 5
  Week 90 | -27.5 [-162.6 to 107.6]
  Week 102: number analyzed (Participants) | 4
  Week 102 | -78.1 [-120.7 to -35.4]
  Week 114: number analyzed (Participants) | 4
  Week 114 | -84.2 [-96.8 to -67.2]
  Week 126: number analyzed (Participants) | 4
  Week 126 | -88.9 [-113.9 to -63.9]
  Week 138: number analyzed (Participants) | 2
  Week 138 | -95.9 [-148.4 to -43.3]
  Week 150: number analyzed (Participants) | 2
  Week 150 | -99.5 [-106.3 to -92.7]
  Week 162: number analyzed (Participants) | 1
  Week 162 | -100.0 [-100.0 to -100.0]
  Week 174: number analyzed (Participants) | 1
  Week 174 | -100.0 [-100.0 to -100.0]
  Week 186: number analyzed (Participants) | 1
  Week 186 | -100.0 [-100.0 to -100.0]
  Week 198: number analyzed (Participants) | 1
  Week 198 | -100.0 [-100.0 to -100.0]

19. Secondary Outcome: Percent Change in Mean Daily Dose of Uveitis-related Systemic Corticosteroids Relative to Week 0 in Participants With Active Uveitis Using Systemic Corticosteroids at Week 0 Over Time
Description: as for outcome 16
Time Frame: Weeks 0, 2, 4, 8, 12, 18, 30, 42, 54, 66, 78, 90, 102, 114, 126, 138, 150, 162, 174, 186, 198, 210, 222, 234, and 246
Population: All participants in the ITT analysis set receiving systemic corticosteroids at Week 0 with evaluable data at a given timepoint.
Measure: Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Adalimumab
Number analyzed (Participants) | 114
percent change from baseline
  Week 2 | -4.6 [-14.2 to 5.0]
  Week 4: number analyzed (Participants) | 112
  Week 4 | -25.0 [-38.6 to -11.4]
  Week 8: number analyzed (Participants) | 112
  Week 8 | -41.7 [-55.0 to -28.4]
  Week 12: number analyzed (Participants) | 107
  Week 12 | -46.3 [-65.0 to -27.7]
  Week 18: number analyzed (Participants) | 106
  Week 18 | -55.1 [-73.1 to -37.1]
  Week 30: number analyzed (Participants) | 102
  Week 30 | -62.8 [-78.1 to -47.5]
  Week 42: number analyzed (Participants) | 96
  Week 42 | -73.4 [-85.0 to -61.9]
  Week 54: number analyzed (Participants) | 93
  Week 54 | -73.2 [-85.3 to -61.0]
  Week 66: number analyzed (Participants) | 87
  Week 66 | -77.1 [-89.3 to -64.9]
  Week 78: number analyzed (Participants) | 84
  Week 78 | -77.3 [-90.2 to -64.4]
  Week 90: number analyzed (Participants) | 80
  Week 90 | -82.1 [-93.3 to -70.9]
  Week 102: number analyzed (Participants) | 76
  Week 102 | -78.8 [-95.7 to -62.0]
  Week 114: number analyzed (Participants) | 72
  Week 114 | -82.0 [-96.8 to -66.9]
  Week 126: number analyzed (Participants) | 65
  Week 126 | -82.8 [-98.6 to -66.9]
  Week 138: number analyzed (Participants) | 62
  Week 138 | -87.8 [-94.2 to -81.4]
  Week 150: number analyzed (Participants) | 57
  Week 150 | -86.9 [-94.5 to -79.2]
  Week 162: number analyzed (Participants) | 55
  Week 162 | -90.7 [-94.9 to -86.4]
  Week 174: number analyzed (Participants) | 52
  Week 174 | -91.4 [-95.8 to -86.9]
  Week 186: number analyzed (Participants) | 47
  Week 186 | -90.3 [-95.9 to -84.7]
  Week 198: number analyzed (Participants) | 42
  Week 198 | -91.0 [-96.6 to -85.5]
  Week 210: number analyzed (Participants) | 38
  Week 210 | -89.9 [-96.8 to -82.9]
  Week 222: number analyzed (Participants) | 30
  Week 222 | -87.1 [-102.0 to -72.2]
  Week 234: number analyzed (Participants) | 20
  Week 234 | -93.8 [-103.8 to -83.9]
  Week 246: number analyzed (Participants) | 18
  Week 246 | -98.3 [-101.3 to -95.4]

20. Secondary Outcome: Percentage of Participants Not Using Systemic Corticosteroids Over Time
Description: Corticosteroid doses were converted into prednisone equivalents. Participants with uveitis-related systemic corticosteroid that could not be converted to prednisone equivalents were excluded. Individual mean daily doses were calculated within the respective visit windows. For Week 0, only uveitis-related systemic corticosteroids at Baseline (Day 1 for all participants) were considered. Baseline was defined as Week 0 for all participants. Data presented for participants not using systemic corticosteroids at each timepoint.
Time Frame: Weeks 0, 2, 4, 8, 12, 18, 30, 42, 54, 66, 78, 90, 102, 114, 126, 138, 150, 162, 174, 186, 198, 210, 222, 234, and 246
Population: All participants in the ITT analysis set with evaluable data at each timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 359
percentage of participants
  Week 0 | 66.3 [61.1 to 71.2]
  Week 2: number analyzed (Participants) | 358
  Week 2 | 58.7 [53.4 to 63.8]
  Week 4: number analyzed (Participants) | 349
  Week 4 | 60.2 [54.8 to 65.3]
  Week 8: number analyzed (Participants) | 339
  Week 8 | 61.9 [56.5 to 67.1]
  Week 12: number analyzed (Participants) | 334
  Week 12 | 64.7 [59.3 to 69.8]
  Week 18: number analyzed (Participants) | 328
  Week 18 | 68.3 [63.0 to 73.3]
  Week 30: number analyzed (Participants) | 312
  Week 30 | 70.2 [64.8 to 75.2]
  Week 42: number analyzed (Participants) | 306
  Week 42 | 70.9 [65.5 to 75.9]
  Week 54: number analyzed (Participants) | 292
  Week 54 | 71.9 [66.4 to 77.0]
  Week 66: number analyzed (Participants) | 275
  Week 66 | 73.1 [67.4 to 78.2]
  Week 78: number analyzed (Participants) | 266
  Week 78 | 75.2 [69.5 to 80.3]
  Week 90: number analyzed (Participants) | 257
  Week 90 | 77.0 [71.4 to 82.0]
  Week 102: number analyzed (Participants) | 239
  Week 102 | 80.8 [75.2 to 85.6]
  Week 114: number analyzed (Participants) | 225
  Week 114 | 83.6 [78.1 to 88.1]
  Week 126: number analyzed (Participants) | 209
  Week 126 | 84.2 [78.5 to 88.9]
  Week 138: number analyzed (Participants) | 190
  Week 138 | 82.1 [75.9 to 87.3]
  Week 150: number analyzed (Participants) | 173
  Week 150 | 81.5 [74.9 to 87.0]
  Week 162: number analyzed (Participants) | 149
  Week 162 | 80.5 [73.3 to 86.6]
  Week 174: number analyzed (Participants) | 136
  Week 174 | 79.4 [71.6 to 85.9]
  Week 186: number analyzed (Participants) | 123
  Week 186 | 80.5 [72.4 to 87.1]
  Week 198: number analyzed (Participants) | 97
  Week 198 | 80.4 [71.1 to 87.8]
  Week 210: number analyzed (Participants) | 82
  Week 210 | 81.7 [71.6 to 89.4]
  Week 222: number analyzed (Participants) | 59
  Week 222 | 86.4 [75.0 to 94.0]
  Week 234: number analyzed (Participants) | 48
  Week 234 | 89.6 [77.3 to 96.5]
  Week 246: number analyzed (Participants) | 34
  Week 246 | 94.1 [80.3 to 99.3]

21. Secondary Outcome: Percentage of Participants Without Worsening of Best Corrected Visual Acuity (BCVA) by ≥15 Letters on Early Treatment Diabetic Retinopathy Study (ETDRS) in Both Eyes Relative to Baseline Over Time Among Participants Who Had Inactive Uveitis at Study Entry
Description: Percentage of participants at each study time point without a worsening of Best Corrected Visual Acuity (BCVA) by ≥15 letters on the Early Treatment Diabetic Retinopathy Study (ETDRS) in both eyes relative to Baseline for participants who had inactive uveitis when they entered the study.
Time Frame: Weeks 2, 4, 8, 12, 18, 30, 42, 54, 66, 78, 90, 102, 114, 126, 138, 150, 162, 174, 186, 198, 210, 222, 234, and 246
Population: All participants in the ITT analysis set with evaluable data at each timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 124
percentage of participants
  Week 2: number analyzed (Participants) | 118
  Week 2 | 100 [96.9 to 100]
  Week 4: number analyzed (Participants) | 108
  Week 4 | 99.1 [94.9 to 100]
  Week 8: number analyzed (Participants) | 113
  Week 8 | 100 [96.8 to 100]
  Week 12: number analyzed (Participants) | 112
  Week 12 | 100 [96.8 to 100]
  Week 18: number analyzed (Participants) | 112
  Week 18 | 100 [96.8 to 100]
  Week 30: number analyzed (Participants) | 112
  Week 30 | 99.1 [95.1 to 100]
  Week 42: number analyzed (Participants) | 112
  Week 42 | 98.2 [93.7 to 99.8]
  Week 54: number analyzed (Participants) | 107
  Week 54 | 97.2 [92.0 to 99.4]
  Week 66: number analyzed (Participants) | 103
  Week 66 | 98.1 [93.2 to 99.8]
  Week 78: number analyzed (Participants) | 99
  Week 78 | 97.0 [91.4 to 99.4]
  Week 90: number analyzed (Participants) | 95
  Week 90 | 98.9 [94.3 to 100]
  Week 102: number analyzed (Participants) | 89
  Week 102 | 97.8 [92.1 to 99.7]
  Week 114: number analyzed (Participants) | 84
  Week 114 | 97.6 [91.7 to 99.7]
  Week 126: number analyzed (Participants) | 76
  Week 126 | 96.1 [88.9 to 99.2]
  Week 138: number analyzed (Participants) | 64
  Week 138 | 96.9 [89.2 to 99.6]
  Week 150: number analyzed (Participants) | 57
  Week 150 | 100 [93.7 to 100]
  Week 162: number analyzed (Participants) | 39
  Week 162 | 100 [91.0 to 100]
  Week 174: number analyzed (Participants) | 34
  Week 174 | 100 [89.7 to 100]
  Week 186: number analyzed (Participants) | 31
  Week 186 | 100 [88.8 to 100]
  Week 198: number analyzed (Participants) | 26
  Week 198 | 100 [86.8 to 100]
  Week 210: number analyzed (Participants) | 16
  Week 210 | 100 [79.4 to 100]
  Week 222: number analyzed (Participants) | 12
  Week 222 | 91.7 [61.5 to 99.8]
  Week 234: number analyzed (Participants) | 9
  Week 234 | 88.9 [51.8 to 99.7]
  Week 246: number analyzed (Participants) | 7
  Week 246 | 85.7 [42.1 to 99.6]

22. Secondary Outcome: Percentage of Participants Without Worsening of BCVA by ≥15 Letters on the ETDRS in Both Eyes Relative to Week 8 Over Time Among Participants With Active Uveitis at Study Entry
Description: Percentage of participants at each study time point without a worsening of BCVA by ≥15 letters on the ETDRS in both eyes relative to Week 8 for participant who had active uveitis when they entered the study.
Time Frame: Weeks 12, 18, 30, 42, 54, 66, 78, 90, 102, 114, 126, 138, 150, 162, 174, 186, 198, 210, 222, 234, and 246
Population: All participants in the ITT analysis set with evaluable data at each timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 222
percentage of participants
  Week 12: number analyzed (Participants) | 219
  Week 12 | 96.8 [93.5 to 98.7]
  Week 18: number analyzed (Participants) | 214
  Week 18 | 96.3 [92.8 to 98.4]
  Week 30: number analyzed (Participants) | 206
  Week 30 | 96.6 [93.1 to 98.6]
  Week 42: number analyzed (Participants) | 196
  Week 42 | 94.9 [90.8 to 97.5]
  Week 54: number analyzed (Participants) | 188
  Week 54 | 94.7 [90.4 to 97.4]
  Week 66: number analyzed (Participants) | 179
  Week 66 | 93.3 [88.6 to 96.5]
  Week 78: number analyzed (Participants) | 172
  Week 78 | 93.6 [88.8 to 96.8]
  Week 90: number analyzed (Participants) | 165
  Week 90 | 96.4 [92.3 to 98.7]
  Week 102: number analyzed (Participants) | 153
  Week 102 | 94.8 [90.0 to 97.7]
  Week 114: number analyzed (Participants) | 146
  Week 114 | 93.8 [88.6 to 97.1]
  Week 126: number analyzed (Participants) | 140
  Week 126 | 95.0 [90.0 to 98.0]
  Week 138: number analyzed (Participants) | 131
  Week 138 | 93.9 [88.3 to 97.3]
  Week 150: number analyzed (Participants) | 123
  Week 150 | 92.7 [86.6 to 96.6]
  Week 162: number analyzed (Participants) | 114
  Week 162 | 93.9 [87.8 to 97.5]
  Week 174: number analyzed (Participants) | 107
  Week 174 | 91.6 [84.6 to 96.1]
  Week 186: number analyzed (Participants) | 96
  Week 186 | 92.7 [85.6 to 97.0]
  Week 198: number analyzed (Participants) | 86
  Week 198 | 95.3 [88.5 to 98.7]
  Week 210: number analyzed (Participants) | 71
  Week 210 | 95.8 [88.1 to 99.1]
  Week 222: number analyzed (Participants) | 58
  Week 222 | 96.6 [88.1 to 99.6]
  Week 234: number analyzed (Participants) | 42
  Week 234 | 95.2 [83.8 to 99.4]
  Week 246: number analyzed (Participants) | 34
  Week 246 | 91.2 [76.3 to 98.1]

23. Secondary Outcome: Mean of Both Eyes of the Logarithm of the Minimum Angle of Resolution (LogMAR) BCVA Over Time
Description: Using corrective lenses based on that visit's refraction testing, participant's BCVA was measured using an ETDRS logMAR chart. On the logMAR scale, 0 is equivalent to 20/20 visual acuity, the range of normal vision is considered to be from -0.2 to 0.1; higher values indicate visual impairment. Data presented includes the mean of both eyes for all participants (active or inactive uveitis) for all study time points.
Time Frame: Weeks 0, 2, 4, 8, 12, 18, 30, 42, 54, 66, 78, 90, 102, 114, 126, 138, 150, 162, 174, 186, 198, 210, 222, 234, and 246
Population: All participants in the ITT analysis set with evaluable data at each study timepoint.
Measure: Mean (Standard Deviation); unit: Log (Mar) BCVA Both Eyes
Arm/Group | Adalimumab
Number analyzed (Participants) | 364
Log (Mar) BCVA Both Eyes
  Week 0 | 0.20 (0.275)
  Week 2: number analyzed (Participants) | 348
  Week 2 | 0.17 (0.265)
  Week 4: number analyzed (Participants) | 325
  Week 4 | 0.15 (0.248)
  Week 8: number analyzed (Participants) | 342
  Week 8 | 0.14 (0.247)
  Week 12: number analyzed (Participants) | 333
  Week 12 | 0.13 (0.244)
  Week 18: number analyzed (Participants) | 329
  Week 18 | 0.12 (0.240)
  Week 30: number analyzed (Participants) | 319
  Week 30 | 0.12 (0.249)
  Week 42: number analyzed (Participants) | 309
  Week 42 | 0.12 (0.227)
  Week 54: number analyzed (Participants) | 296
  Week 54 | 0.11 (0.238)
  Week 66: number analyzed (Participants) | 284
  Week 66 | 0.11 (0.241)
  Week 78: number analyzed (Participants) | 272
  Week 78 | 0.11 (0.238)
  Week 90: number analyzed (Participants) | 261
  Week 90 | 0.09 (0.214)
  Week 102: number analyzed (Participants) | 244
  Week 102 | 0.09 (0.219)
  Week 114: number analyzed (Participants) | 231
  Week 114 | 0.09 (0.233)
  Week 126: number analyzed (Participants) | 217
  Week 126 | 0.09 (0.231)
  Week 138: number analyzed (Participants) | 197
  Week 138 | 0.09 (0.224)
  Week 150: number analyzed (Participants) | 181
  Week 150 | 0.10 (0.255)
  Week 162: number analyzed (Participants) | 154
  Week 162 | 0.09 (0.249)
  Week 174: number analyzed (Participants) | 142
  Week 174 | 0.09 (0.261)
  Week 186: number analyzed (Participants) | 128
  Week 186 | 0.09 (0.244)
  Week 198: number analyzed (Participants) | 113
  Week 198 | 0.07 (0.205)
  Week 210: number analyzed (Participants) | 88
  Week 210 | 0.07 (0.211)
  Week 222: number analyzed (Participants) | 71
  Week 222 | 0.07 (0.218)
  Week 234: number analyzed (Participants) | 51
  Week 234 | 0.07 (0.222)
  Week 246: number analyzed (Participants) | 41
  Week 246 | 0.08 (0.217)

24. Other Pre Specified Outcome: Percent Change in Left Eye in Central Retinal Thickness (1 mm Subfield) From Baseline to Each Study Time Point Relative to Baseline for Participants Who Had Inactive Uveitis at Study Entry Over Time
Description: Central retinal thickness was measured using optical coherence tomography (OCT) and assessed by a central reader. Percent change in left eye from baseline (Week 0) to each study time point relative to baseline for participants who had inactive uveitis at study entry is presented.
Time Frame: Baseline (Week 0) and Weeks 2, 4, 8, 12, 18, 30, 42, 54, 66, 78, 90, 102, 114, 126, 138, 150, 162, 174, 186, 198, 210, 222, 234, and 246
Population: All participants in the ITT analysis set with evaluable data at each timepoint.
Measure: Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Adalimumab
Number analyzed (Participants) | 111
percent change from baseline
  Week 2 | 0.3 [-1.41 to 1.97]
  Week 4: number analyzed (Participants) | 100
  Week 4 | -0.2 [-2.03 to 1.56]
  Week 8: number analyzed (Participants) | 106
  Week 8 | -0.7 [-2.07 to 0.72]
  Week 12: number analyzed (Participants) | 105
  Week 12 | -1.0 [-2.27 to 0.23]
  Week 18: number analyzed (Participants) | 105
  Week 18 | -0.5 [-2.02 to 1.07]
  Week 30: number analyzed (Participants) | 104
  Week 30 | -1.9 [-3.25 to -0.60]
  Week 42: number analyzed (Participants) | 103
  Week 42 | -1.3 [-2.83 to 0.17]
  Week 54: number analyzed (Participants) | 101
  Week 54 | -2.1 [-3.90 to -0.22]
  Week 66: number analyzed (Participants) | 96
  Week 66 | -1.9 [-3.95 to 0.11]
  Week 78: number analyzed (Participants) | 88
  Week 78 | -1.4 [-4.54 to 1.70]
  Week 90: number analyzed (Participants) | 85
  Week 90 | -2.9 [-4.51 to -1.22]
  Week 102: number analyzed (Participants) | 82
  Week 102 | -3.1 [-4.95 to -1.34]
  Week 114: number analyzed (Participants) | 75
  Week 114 | -2.8 [-4.44 to -1.14]
  Week 126: number analyzed (Participants) | 67
  Week 126 | -3.7 [-5.66 to -1.68]
  Week 138: number analyzed (Participants) | 58
  Week 138 | -3.4 [-5.38 to -1.46]
  Week 150: number analyzed (Participants) | 52
  Week 150 | -3.5 [-5.48 to -1.58]
  Week 162: number analyzed (Participants) | 32
  Week 162 | -3.3 [-6.25 to -0.29]
  Week 174: number analyzed (Participants) | 29
  Week 174 | -3.0 [-5.45 to -0.52]
  Week 186: number analyzed (Participants) | 27
  Week 186 | -3.8 [-6.69 to -1.00]
  Week 198: number analyzed (Participants) | 23
  Week 198 | -3.2 [-5.99 to -0.35]
  Week 210: number analyzed (Participants) | 13
  Week 210 | -5.2 [-10.23 to -0.17]
  Week 222: number analyzed (Participants) | 10
  Week 222 | -4.6 [-11.17 to 1.93]
  Week 234: number analyzed (Participants) | 8
  Week 234 | -3.6 [-13.06 to 5.77]
  Week 246: number analyzed (Participants) | 6
  Week 246 | -3.4 [-14.83 to 7.93]

25. Other Pre Specified Outcome: Percent Change in Right Eye in Central Retinal Thickness (1 mm Subfield) From Baseline to Each Study Time Point Relative to Baseline for Participants Who Had Inactive Uveitis at Study Entry Over Time
Description: Central retinal thickness was measured using optical coherence tomography (OCT) and assessed by a central reader. Percent change in right eye from baseline (Week 0) to each study time point relative to baseline for participants who had inactive uveitis at study entry is presented.
Time Frame: as for outcome 24
Population: All participants in the ITT analysis set with evaluable data at each timepoint.
Measure: Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Adalimumab
Number analyzed (Participants) | 109
percent change from baseline
  Week 2 | -0.2 [-1.92 to 1.45]
  Week 4: number analyzed (Participants) | 99
  Week 4 | -0.8 [-2.99 to 1.39]
  Week 8: number analyzed (Participants) | 104
  Week 8 | -1.5 [-3.19 to 0.25]
  Week 12: number analyzed (Participants) | 103
  Week 12 | -1.0 [-2.76 to 0.66]
  Week 18: number analyzed (Participants) | 103
  Week 18 | -0.4 [-2.73 to 1.84]
  Week 30: number analyzed (Participants) | 102
  Week 30 | -2.8 [-4.78 to -0.86]
  Week 42: number analyzed (Participants) | 101
  Week 42 | -2.2 [-4.31 to -0.15]
  Week 54: number analyzed (Participants) | 99
  Week 54 | -3.7 [-6.00 to -1.44]
  Week 66: number analyzed (Participants) | 94
  Week 66 | -3.3 [-5.66 to -0.97]
  Week 78: number analyzed (Participants) | 86
  Week 78 | -3.9 [-6.36 to -1.38]
  Week 90: number analyzed (Participants) | 83
  Week 90 | -3.8 [-6.47 to -1.08]
  Week 102: number analyzed (Participants) | 80
  Week 102 | -5.3 [-7.99 to -2.67]
  Week 114: number analyzed (Participants) | 73
  Week 114 | -5.6 [-8.65 to -2.53]
  Week 126: number analyzed (Participants) | 65
  Week 126 | -5.4 [-8.57 to -2.21]
  Week 138: number analyzed (Participants) | 56
  Week 138 | -4.7 [-7.75 to -1.72]
  Week 150: number analyzed (Participants) | 51
  Week 150 | -2.1 [-9.07 to 4.90]
  Week 162: number analyzed (Participants) | 32
  Week 162 | -2.9 [-6.06 to 0.36]
  Week 174: number analyzed (Participants) | 29
  Week 174 | -2.7 [-5.88 to 0.56]
  Week 186: number analyzed (Participants) | 27
  Week 186 | -2.0 [-5.49 to 1.46]
  Week 198: number analyzed (Participants) | 23
  Week 198 | -1.2 [-5.91 to 3.48]
  Week 210: number analyzed (Participants) | 13
  Week 210 | -2.3 [-6.35 to 1.66]
  Week 222: number analyzed (Participants) | 10
  Week 222 | -1.7 [-4.76 to 1.44]
  Week 234: number analyzed (Participants) | 8
  Week 234 | -1.3 [-6.32 to 3.78]
  Week 246: number analyzed (Participants) | 6
  Week 246 | 1.6 [-0.78 to 3.93]

26. Other Pre Specified Outcome: Percent Change in Left Eye of Central Retinal Thickness (1 mm Subfield) at Each Study Time Point Relative to Week 8 for Participants Who Had Active Uveitis at Study Entry Over Time
Description: Central retinal thickness was measured using OCT and assessed by a central reader. Percent change in left eye at each study time point relative to Week 8 (baseline) for participants who had active uveitis at study entry is presented.
Time Frame: Baseline (Week 8) and Weeks 12, 18, 30, 42, 54, 66, 78, 90, 102, 114, 126, 138, 150, 162, 174, 186, 198, 210, 222, 234, and 246
Population: All participants in the ITT analysis set with evaluable data at each timepoint.
Measure: Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Adalimumab
Number analyzed (Participants) | 206
percent change from baseline
  Week 12 | 1.0 [-0.50 to 2.42]
  Week 18: number analyzed (Participants) | 201
  Week 18 | -0.3 [-2.36 to 1.71]
  Week 30: number analyzed (Participants) | 194
  Week 30 | -2.4 [-4.24 to -0.55]
  Week 42: number analyzed (Participants) | 183
  Week 42 | -2.8 [-4.62 to -1.00]
  Week 54: number analyzed (Participants) | 177
  Week 54 | -3.2 [-5.52 to -0.90]
  Week 66: number analyzed (Participants) | 166
  Week 66 | -2.3 [-4.52 to 0.01]
  Week 78: number analyzed (Participants) | 161
  Week 78 | -3.5 [-5.99 to -1.02]
  Week 90: number analyzed (Participants) | 150
  Week 90 | -4.8 [-7.19 to -2.42]
  Week 102: number analyzed (Participants) | 142
  Week 102 | -5.3 [-7.41 to -3.10]
  Week 114: number analyzed (Participants) | 126
  Week 114 | -6.6 [-9.15 to -3.95]
  Week 126: number analyzed (Participants) | 124
  Week 126 | -5.3 [-8.66 to -1.92]
  Week 138: number analyzed (Participants) | 118
  Week 138 | -7.0 [-9.96 to -3.99]
  Week 150: number analyzed (Participants) | 109
  Week 150 | -7.3 [-10.22 to -4.48]
  Week 162: number analyzed (Participants) | 104
  Week 162 | -7.5 [-11.31 to -3.72]
  Week 174: number analyzed (Participants) | 92
  Week 174 | -9.5 [-13.20 to -5.81]
  Week 186: number analyzed (Participants) | 83
  Week 186 | -7.6 [-10.21 to -4.93]
  Week 198: number analyzed (Participants) | 74
  Week 198 | -8.4 [-11.84 to -4.99]
  Week 210: number analyzed (Participants) | 67
  Week 210 | -6.6 [-10.40 to -2.74]
  Week 222: number analyzed (Participants) | 53
  Week 222 | -9.3 [-13.42 to -5.17]
  Week 234: number analyzed (Participants) | 39
  Week 234 | -8.2 [-11.85 to -4.46]
  Week 246: number analyzed (Participants) | 32
  Week 246 | -9.1 [-13.41 to -4.82]

27. Other Pre Specified Outcome: Percent Change in Right Eye of Central Retinal Thickness (1 mm Subfield) at Each Study Time Point Relative to Week 8 for Participants Who Had Active Uveitis at Study Entry Over Time
Description: Central retinal thickness was measured using OCT and assessed by a central reader. Percent change in right eye at each study time point relative to Week 8 (baseline) for participants who had active uveitis at study entry is presented.
Time Frame: as for outcome 26
Population: All participants in the ITT analysis set with evaluable data at each timepoint.
Measure: Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Adalimumab
Number analyzed (Participants) | 205
percent change from baseline
  Week 12 | 0.4 [-1.58 to 2.47]
  Week 18: number analyzed (Participants) | 202
  Week 18 | -0.7 [-2.71 to 1.30]
  Week 30: number analyzed (Participants) | 194
  Week 30 | -0.7 [-3.36 to 1.90]
  Week 42: number analyzed (Participants) | 183
  Week 42 | -2.4 [-4.85 to 0.05]
  Week 54: number analyzed (Participants) | 176
  Week 54 | -2.4 [-5.25 to 0.36]
  Week 66: number analyzed (Participants) | 167
  Week 66 | -1.3 [-4.81 to 2.27]
  Week 78: number analyzed (Participants) | 160
  Week 78 | -2.1 [-5.61 to 1.50]
  Week 90: number analyzed (Participants) | 149
  Week 90 | -3.6 [-6.44 to -0.76]
  Week 102: number analyzed (Participants) | 142
  Week 102 | -3.4 [-6.98 to 0.13]
  Week 114: number analyzed (Participants) | 125
  Week 114 | -2.2 [-6.18 to 1.81]
  Week 126: number analyzed (Participants) | 124
  Week 126 | -3.5 [-7.43 to 0.47]
  Week 138: number analyzed (Participants) | 118
  Week 138 | -4.6 [-8.22 to -0.92]
  Week 150: number analyzed (Participants) | 109
  Week 150 | -6.5 [-9.81 to -3.15]
  Week 162: number analyzed (Participants) | 104
  Week 162 | -4.8 [-8.91 to -0.75]
  Week 174: number analyzed (Participants) | 93
  Week 174 | -5.4 [-9.46 to -1.27]
  Week 186: number analyzed (Participants) | 83
  Week 186 | -7.9 [-12.74 to -3.03]
  Week 198: number analyzed (Participants) | 75
  Week 198 | -8.2 [-12.30 to -4.13]
  Week 210: number analyzed (Participants) | 67
  Week 210 | -6.6 [-10.76 to -2.43]
  Week 222: number analyzed (Participants) | 52
  Week 222 | -9.7 [-13.24 to -6.19]
  Week 234: number analyzed (Participants) | 39
  Week 234 | -9.7 [-14.24 to -5.07]
  Week 246: number analyzed (Participants) | 32
  Week 246 | -9.9 [-15.43 to -4.35]

28. Other Pre Specified Outcome: Percentage of Participants With Grade ≤0.5+ in Anterior Chamber (AC) Cells in Both Eyes on Slit Lamp Exam According to Standardization of Uveitis Nomenclature (SUN) Criteria Over Time
Description: Slit lamp examinations were conducted at each visit to assess AC cell count. The number of AC cells observed within a 1 mm * 1 mm slit beam was used to determine the grade according to the Standardization of Uveitis Nomenclature (SUN) criteria: Grade 0: ˂ 1 cell; Grade 0.5+: 1 - 5 cells; Grade 1+: 6 - 15 cells; Grade 2+: 16 - 25 cells; Grade 3+: 26 - 50 cells; and Grade 4+: ≥ 50 cells.
Time Frame: Weeks 0, 2, 4, 8, 12, 18, 30, 42, 54, 66, 78, 90, 102, 114, 126, 138, 150, 162, 174, 186, 198, 210, 222, 234, and 246
Population: All participants in the ITT analysis set with evaluable data at each timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 364
percentage of participants
  Week 0 | 65.4 [60.3 to 70.3]
  Week 2: number analyzed (Participants) | 348
  Week 2 | 85.9 [81.8 to 89.4]
  Week 4: number analyzed (Participants) | 323
  Week 4 | 90.4 [86.7 to 93.4]
  Week 8: number analyzed (Participants) | 343
  Week 8 | 91.5 [88.1 to 94.3]
  Week 12: number analyzed (Participants) | 333
  Week 12 | 91.3 [87.7 to 94.1]
  Week 18: number analyzed (Participants) | 330
  Week 18 | 90.9 [87.3 to 93.8]
  Week 30: number analyzed (Participants) | 319
  Week 30 | 94.7 [91.6 to 96.9]
  Week 42: number analyzed (Participants) | 310
  Week 42 | 92.3 [88.7 to 95.0]
  Week 54: number analyzed (Participants) | 296
  Week 54 | 92.9 [89.4 to 95.6]
  Week 66: number analyzed (Participants) | 284
  Week 66 | 95.1 [91.9 to 97.3]
  Week 78: number analyzed (Participants) | 272
  Week 78 | 93.0 [89.3 to 95.7]
  Week 90: number analyzed (Participants) | 261
  Week 90 | 94.3 [90.7 to 96.7]
  Week 102: number analyzed (Participants) | 245
  Week 102 | 93.5 [89.6 to 96.2]
  Week 114: number analyzed (Participants) | 231
  Week 114 | 93.5 [89.5 to 96.3]
  Week 126: number analyzed (Participants) | 217
  Week 126 | 94.0 [90.0 to 96.8]
  Week 138: number analyzed (Participants) | 197
  Week 138 | 93.4 [89.0 to 96.4]
  Week 150: number analyzed (Participants) | 181
  Week 150 | 94.5 [90.1 to 97.3]
  Week 162: number analyzed (Participants) | 154
  Week 162 | 95.5 [90.9 to 98.2]
  Week 174: number analyzed (Participants) | 142
  Week 174 | 94.4 [89.2 to 97.5]
  Week 186: number analyzed (Participants) | 128
  Week 186 | 96.1 [91.1 to 98.7]
  Week 198: number analyzed (Participants) | 113
  Week 198 | 94.7 [88.8 to 98.0]
  Week 210: number analyzed (Participants) | 89
  Week 210 | 96.6 [90.5 to 99.3]
  Week 222: number analyzed (Participants) | 71
  Week 222 | 98.6 [92.4 to 100]
  Week 234: number analyzed (Participants) | 51
  Week 234 | 100 [93.0 to 100]
  Week 246: number analyzed (Participants) | 42
  Week 246 | 95.2 [83.8 to 99.4]

29. Other Pre Specified Outcome: Percentage of Participants Achieving a ≥50% Reduction in Immunosuppression Load Relative to Baseline Over Time Among Participants With Inactive Uveitis at Study Entry
Description: Immunosuppression load was assessed using a weighted semiquantitative scale, applying grades ranging from 0 to 9 for each immunosuppressive agent on a scale for the total daily dose in milligrams per kilogram per day or per week if dosed weekly. A higher score indicating a higher immunosuppression load and a lower or decreased score indicated improvement or less need for immunosuppressive therapy. The grading scheme was used to accommodate the simultaneous use of multiple agents and provided a combined, single numeric score for the total immunosuppression load per unit body weight per day at each visit. For participants receiving multiple medications, the sum of the grading scores for each drug was used to calculate a total immunosuppression score at each visit. Data not presented after Week 234 as no participants remained on study as of Week 234.
Time Frame: Weeks 2, 4, 8, 12, 18, 30, 42, 54, 66, 78, 90, 102, 114, 126, 138, 150, 162, 174, 186, 198, 210, 222, and 234
Population: All participants in the ITT analysis set with an immunosuppression load greater than 0 at baseline (Week 0) with evaluable data at each timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 55
percentage of participants
  Week 2 | 3.6 [0.4 to 12.5]
  Week 4 | 9.1 [3.0 to 20.0]
  Week 8: number analyzed (Participants) | 52
  Week 8 | 17.3 [8.2 to 30.3]
  Week 12: number analyzed (Participants) | 52
  Week 12 | 17.3 [8.2 to 30.3]
  Week 18: number analyzed (Participants) | 51
  Week 18 | 21.6 [11.3 to 35.3]
  Week 30: number analyzed (Participants) | 49
  Week 30 | 24.5 [13.3 to 38.9]
  Week 42: number analyzed (Participants) | 48
  Week 42 | 22.9 [12.0 to 37.3]
  Week 54: number analyzed (Participants) | 45
  Week 54 | 17.8 [8.0 to 32.1]
  Week 66: number analyzed (Participants) | 40
  Week 66 | 15.0 [5.7 to 29.8]
  Week 78: number analyzed (Participants) | 40
  Week 78 | 15.0 [5.7 to 29.8]
  Week 90: number analyzed (Participants) | 37
  Week 90 | 13.5 [4.5 to 28.8]
  Week 102: number analyzed (Participants) | 34
  Week 102 | 14.7 [5.0 to 31.1]
  Week 114: number analyzed (Participants) | 32
  Week 114 | 25.0 [11.5 to 43.4]
  Week 126: number analyzed (Participants) | 28
  Week 126 | 25.0 [10.7 to 44.9]
  Week 138: number analyzed (Participants) | 24
  Week 138 | 25.0 [9.8 to 46.7]
  Week 150: number analyzed (Participants) | 21
  Week 150 | 23.8 [8.2 to 47.2]
  Week 162: number analyzed (Participants) | 16
  Week 162 | 18.8 [4.0 to 45.6]
  Week 174: number analyzed (Participants) | 16
  Week 174 | 12.5 [1.6 to 38.3]
  Week 186: number analyzed (Participants) | 16
  Week 186 | 12.5 [1.6 to 38.3]
  Week 198: number analyzed (Participants) | 10
  Week 198 | 0 [0 to 0]
  Week 210: number analyzed (Participants) | 8
  Week 210 | 12.5 [0.3 to 52.7]
  Week 222: number analyzed (Participants) | 4
  Week 222 | 25.0 [0.6 to 80.6]
  Week 234: number analyzed (Participants) | 4
  Week 234 | 50.0 [6.8 to 93.2]

30. Other Pre Specified Outcome: Percentage of Participants Achieving a ≥50% Reduction in Immunosuppression Load Relative to Week 8 Over Time Among Participants With Active Uveitis at Study Entry
Description: Immunosuppression load was assessed using a weighted semiquantitative scale, applying grades ranging from 0 to 9 for each immunosuppressive agent on a scale for the total daily dose in milligrams per kilogram per day or per week if dosed weekly. A higher score indicating a higher immunosuppression load and a lower or decreased score indicated improvement or less need for immunosuppressive therapy. The grading scheme was used to accommodate the simultaneous use of multiple agents and provided a combined, single numeric score for the total immunosuppression load per unit body weight per day at each visit. For participants receiving multiple medications, the sum of the grading scores for each drug was used to calculate a total immunosuppression score at each visit.
Time Frame: Weeks 12, 18, 30, 42, 54, 66, 78, 90, 102, 114, 126, 138, 150, 162, 174, 186, 198, 210, 222, 234, and 246
Population: All participants in the ITT analysis set with an immunosuppression load greater than 0 at baseline (Week 8) with evaluable data at each timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 140
percentage of participants
  Week 12 | 17.1 [11.3 to 24.4]
  Week 18: number analyzed (Participants) | 136
  Week 18 | 27.2 [19.9 to 35.5]
  Week 30: number analyzed (Participants) | 128
  Week 30 | 33.6 [25.5 to 42.5]
  Week 42: number analyzed (Participants) | 125
  Week 42 | 41.6 [32.9 to 50.8]
  Week 54: number analyzed (Participants) | 119
  Week 54 | 44.5 [35.4 to 53.9]
  Week 66: number analyzed (Participants) | 113
  Week 66 | 48.7 [39.2 to 58.3]
  Week 78: number analyzed (Participants) | 109
  Week 78 | 48.6 [38.9 to 58.4]
  Week 90: number analyzed (Participants) | 106
  Week 90 | 53.8 [43.8 to 63.5]
  Week 102: number analyzed (Participants) | 98
  Week 102 | 54.1 [43.7 to 64.2]
  Week 114: number analyzed (Participants) | 90
  Week 114 | 51.1 [40.3 to 61.8]
  Week 126: number analyzed (Participants) | 87
  Week 126 | 52.9 [41.9 to 63.7]
  Week 138: number analyzed (Participants) | 80
  Week 138 | 52.5 [41.0 to 63.8]
  Week 150: number analyzed (Participants) | 76
  Week 150 | 53.9 [42.1 to 65.5]
  Week 162: number analyzed (Participants) | 71
  Week 162 | 53.5 [41.3 to 65.5]
  Week 174: number analyzed (Participants) | 63
  Week 174 | 55.6 [42.5 to 68.1]
  Week 186: number analyzed (Participants) | 59
  Week 186 | 55.9 [42.4 to 68.8]
  Week 198: number analyzed (Participants) | 50
  Week 198 | 52.0 [37.4 to 66.3]
  Week 210: number analyzed (Participants) | 41
  Week 210 | 51.2 [35.1 to 67.1]
  Week 222: number analyzed (Participants) | 31
  Week 222 | 54.8 [36.0 to 72.7]
  Week 234: number analyzed (Participants) | 23
  Week 234 | 56.5 [34.5 to 76.8]
  Week 246: number analyzed (Participants) | 19
  Week 246 | 63.2 [38.4 to 83.7]

31. Other Pre Specified Outcome: Percentage of Participants With No New Active, Inflammatory Chorioretinal or Inflammatory Retinal Vascular Lesion in Both Eyes Relative to Baseline Over Time Among Participants With Inactive Uveitis at Study Entry
Description: Percentage of participants at each study time point with no new active, inflammatory chorioretinal or inflammatory retinal vascular lesion in both eyes relative to Baseline for participants who had inactive uveitis when they entered the study.
Time Frame: Weeks 2, 4, 8, 12, 18, 30, 42, 54, 66, 78, 90, 102, 114, 126, 138, 150, 162, 174, 186, 198, 210, 222, 234, and 246
Population: All participants in the ITT analysis set that had evaluable data at each timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 124
percentage of participants
  Week 2: number analyzed (Participants) | 118
  Week 2 | 100 [96.9 to 100]
  Week 4: number analyzed (Participants) | 107
  Week 4 | 99.1 [94.9 to 100]
  Week 8: number analyzed (Participants) | 113
  Week 8 | 100 [96.8 to 100]
  Week 12: number analyzed (Participants) | 112
  Week 12 | 100 [96.8 to 100]
  Week 18: number analyzed (Participants) | 112
  Week 18 | 98.2 [93.7 to 99.8]
  Week 30: number analyzed (Participants) | 112
  Week 30 | 100 [96.8 to 100]
  Week 42: number analyzed (Participants) | 112
  Week 42 | 98.2 [93.7 to 99.8]
  Week 54: number analyzed (Participants) | 107
  Week 54 | 99.1 [94.9 to 100]
  Week 66: number analyzed (Participants) | 103
  Week 66 | 100 [96.5 to 100]
  Week 78: number analyzed (Participants) | 99
  Week 78 | 100 [96.3 to 100]
  Week 90: number analyzed (Participants) | 95
  Week 90 | 98.9 [94.3 to 100]
  Week 102: number analyzed (Participants) | 89
  Week 102 | 98.9 [93.9 to 100]
  Week 114: number analyzed (Participants) | 84
  Week 114 | 100 [95.7 to 100]
  Week 126: number analyzed (Participants) | 75
  Week 126 | 100 [95.2 to 100]
  Week 138: number analyzed (Participants) | 64
  Week 138 | 98.4 [91.6 to 100]
  Week 150: number analyzed (Participants) | 57
  Week 150 | 96.5 [87.9 to 99.6]
  Week 162: number analyzed (Participants) | 39
  Week 162 | 97.4 [86.5 to 99.9]
  Week 174: number analyzed (Participants) | 34
  Week 174 | 100 [89.7 to 100]
  Week 186: number analyzed (Participants) | 31
  Week 186 | 100 [88.8 to 100]
  Week 198: number analyzed (Participants) | 26
  Week 198 | 100 [86.8 to 100]
  Week 210: number analyzed (Participants) | 16
  Week 210 | 100 [79.4 to 100]
  Week 222: number analyzed (Participants) | 12
  Week 222 | 100 [73.5 to 100]
  Week 234: number analyzed (Participants) | 9
  Week 234 | 100 [66.4 to 100]
  Week 246: number analyzed (Participants) | 7
  Week 246 | 100 [59.0 to 100]

32. Other Pre Specified Outcome: Percentage of Participants With No New Active, Inflammatory Chorioretinal or Inflammatory Retinal Vascular Lesion in Both Eyes Relative to Week 8 Over Time Among Participants With Active Uveitis at Study Entry
Description: Percentage of participants at each study time point with no new active, inflammatory chorioretinal or inflammatory retinal vascular lesion in both eyes relative to Week 8 for participants who had active uveitis when they entered the study.
Time Frame: Weeks 12, 18, 30, 42, 54, 66, 78, 90, 102, 114, 126, 138, 150, 162, 174, 186, 198, 210, 222, 234, and 246
Population: All participants in the ITT analysis set with evaluable data at each timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 225
percentage of participants
  Week 12: number analyzed (Participants) | 221
  Week 12 | 97.7 [94.8 to 99.3]
  Week 18: number analyzed (Participants) | 218
  Week 18 | 99.1 [96.7 to 99.9]
  Week 30: number analyzed (Participants) | 207
  Week 30 | 97.1 [93.8 to 98.9]
  Week 42: number analyzed (Participants) | 198
  Week 42 | 99.0 [96.4 to 99.9]
  Week 54: number analyzed (Participants) | 188
  Week 54 | 98.9 [96.2 to 99.9]
  Week 66: number analyzed (Participants) | 181
  Week 66 | 98.3 [95.2 to 99.7]
  Week 78: number analyzed (Participants) | 173
  Week 78 | 97.7 [94.2 to 99.4]
  Week 90: number analyzed (Participants) | 166
  Week 90 | 97.6 [93.9 to 99.3]
  Week 102: number analyzed (Participants) | 156
  Week 102 | 99.4 [96.5 to 100]
  Week 114: number analyzed (Participants) | 147
  Week 114 | 97.3 [93.2 to 99.3]
  Week 126: number analyzed (Participants) | 140
  Week 126 | 99.3 [96.1 to 100]
  Week 138: number analyzed (Participants) | 132
  Week 138 | 100 [97.2 to 100]
  Week 150: number analyzed (Participants) | 123
  Week 150 | 96.7 [91.9 to 99.1]
  Week 162: number analyzed (Participants) | 115
  Week 162 | 97.4 [92.6 to 99.5]
  Week 174: number analyzed (Participants) | 108
  Week 174 | 100 [96.6 to 100]
  Week 186: number analyzed (Participants) | 97
  Week 186 | 99.0 [94.4 to 100]
  Week 198: number analyzed (Participants) | 87
  Week 198 | 100 [95.8 to 100]
  Week 210: number analyzed (Participants) | 73
  Week 210 | 100 [95.1 to 100]
  Week 222: number analyzed (Participants) | 59
  Week 222 | 100 [93.9 to 100]
  Week 234: number analyzed (Participants) | 42
  Week 234 | 100 [91.6 to 100]
  Week 246: number analyzed (Participants) | 35
  Week 246 | 100 [90.0 to 100]

33. Other Pre Specified Outcome: Percentage of Participants With Grade ≤0.5+ in VH in Both Eyes on Indirect Ophthalmoscopy According to NEI/SUN Criteria Over Time
Description: Vitreous haze was measured using dilated indirect ophthalmoscopy (DIO) and assessed by the Investigator according to NEI and SUN criteria:
  Grade 0: No evident vitreous haze; Grade 0.5+: Slight blurring of the optic disc margin because of the haze; normal striations and reflex of the nerve fiber layer cannot be visualized; Grade 1+: Permits a better definition of both the optic nerve head and the retinal vessels (compared to higher grades); Grade 2+: Permits better visualization of the retinal vessels (compared to higher grades); Grade 3+: Permits the observer to see the optic nerve head, but the borders are quite blurry; Grade 4+: Optic nerve head is obscured.
Time Frame: Weeks 0, 2, 4, 8, 12, 18, 30, 42, 54, 66, 78, 90, 102, 114, 126, 138, 150, 162, 174, 186, 198, 210, 222, 234, and 246
Population: All participants in the ITT analysis set with evaluable data at each timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 364
percentage of participants
  Week 0 | 58.0 [52.7 to 63.1]
  Week 2: number analyzed (Participants) | 348
  Week 2 | 75.6 [70.7 to 80.0]
  Week 4: number analyzed (Participants) | 323
  Week 4 | 77.7 [72.8 to 82.1]
  Week 8: number analyzed (Participants) | 342
  Week 8 | 84.2 [79.9 to 87.9]
  Week 12: number analyzed (Participants) | 333
  Week 12 | 84.4 [80.0 to 88.1]
  Week 18: number analyzed (Participants) | 330
  Week 18 | 87.3 [83.2 to 90.7]
  Week 30: number analyzed (Participants) | 319
  Week 30 | 87.1 [83.0 to 90.6]
  Week 42: number analyzed (Participants) | 310
  Week 42 | 90.3 [86.5 to 93.4]
  Week 54: number analyzed (Participants) | 295
  Week 54 | 89.5 [85.4 to 92.7]
  Week 66: number analyzed (Participants) | 283
  Week 66 | 92.2 [88.5 to 95.1]
  Week 78: number analyzed (Participants) | 270
  Week 78 | 93.3 [89.7 to 96.0]
  Week 90: number analyzed (Participants) | 261
  Week 90 | 93.5 [89.8 to 96.2]
  Week 102: number analyzed (Participants) | 245
  Week 102 | 93.9 [90.1 to 96.5]
  Week 114: number analyzed (Participants) | 231
  Week 114 | 93.1 [89.0 to 96.0]
  Week 126: number analyzed (Participants) | 215
  Week 126 | 94.9 [91.0 to 97.4]
  Week 138: number analyzed (Participants) | 196
  Week 138 | 95.4 [91.5 to 97.9]
  Week 150: number analyzed (Participants) | 180
  Week 150 | 92.2 [87.3 to 95.7]
  Week 162: number analyzed (Participants) | 154
  Week 162 | 91.6 [86.0 to 95.4]
  Week 174: number analyzed (Participants) | 142
  Week 174 | 92.3 [86.6 to 96.1]
  Week 186: number analyzed (Participants) | 128
  Week 186 | 96.1 [91.1 to 98.7]
  Week 198: number analyzed (Participants) | 113
  Week 198 | 93.8 [87.7 to 97.5]
  Week 210: number analyzed (Participants) | 88
  Week 210 | 92.0 [84.3 to 96.7]
  Week 222: number analyzed (Participants) | 70
  Week 222 | 95.7 [88.0 to 99.1]
  Week 234: number analyzed (Participants) | 51
  Week 234 | 96.1 [86.5 to 99.5]
  Week 246: number analyzed (Participants) | 42
  Week 246 | 97.6 [87.4 to 99.9]

34. Other Pre Specified Outcome: Change in National Eye Institute (NEI) Visual Functioning Questionnaire (VFQ-25) Score at Each Study Time Point Relative to Baseline for Participants Who Had Inactive Uveitis at Study Entry Over Time
Description: The National Eye Institute (NEI) Visual Functioning Questionnaire (VFQ-25) is an ocular disease-specific survey that measures the influence of visual disability and visual symptoms on generic health domains such as emotional well-being and social functioning, in addition to task-oriented domains related to daily visual functioning.The VFQ-25 consists of a base set of 25 vision-targeted questions plus an additional single-item general health rating question. The overall composite score ranges from 0 to 100, where higher scores or increases in score indicate better vision-related functioning. Baseline was defined as Week 0 for participants with inactive uveitis.
Time Frame: Weeks 0, 8, 18, 30, 42, 54, 66, 78, 90, 102, 114, 126, 138, 150, 162, 174, 186, 198, 210, 222, 234, and 246
Population: All participants in the ITT analysis set with evaluable data at each timepoint.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 122
score on a scale
  Week 0 | 84.77 [81.93 to 87.62]
  Week 8: number analyzed (Participants) | 111
  Week 8 | 84.37 [81.37 to 87.37]
  Week 18: number analyzed (Participants) | 112
  Week 18 | 85.21 [82.30 to 88.13]
  Week 30: number analyzed (Participants) | 111
  Week 30 | 84.75 [81.91 to 87.59]
  Week 42: number analyzed (Participants) | 111
  Week 42 | 84.41 [81.29 to 87.53]
  Week 54: number analyzed (Participants) | 105
  Week 54 | 84.87 [81.82 to 87.91]
  Week 66: number analyzed (Participants) | 103
  Week 66 | 84.09 [80.97 to 87.21]
  Week 78: number analyzed (Participants) | 99
  Week 78 | 83.59 [80.33 to 86.85]
  Week 90: number analyzed (Participants) | 95
  Week 90 | 83.66 [80.18 to 87.15]
  Week 102: number analyzed (Participants) | 89
  Week 102 | 84.19 [80.62 to 87.76]
  Week 114: number analyzed (Participants) | 83
  Week 114 | 84.09 [80.40 to 87.78]
  Week 126: number analyzed (Participants) | 76
  Week 126 | 84.44 [80.59 to 88.28]
  Week 138: number analyzed (Participants) | 64
  Week 138 | 84.85 [80.56 to 89.14]
  Week 150: number analyzed (Participants) | 57
  Week 150 | 83.90 [78.95 to 88.85]
  Week 162: number analyzed (Participants) | 39
  Week 162 | 86.60 [81.31 to 91.90]
  Week 174: number analyzed (Participants) | 34
  Week 174 | 87.25 [81.51 to 92.99]
  Week 186: number analyzed (Participants) | 31
  Week 186 | 87.25 [81.43 to 93.06]
  Week 198: number analyzed (Participants) | 26
  Week 198 | 85.30 [78.35 to 92.26]
  Week 210: number analyzed (Participants) | 16
  Week 210 | 85.71 [76.61 to 94.82]
  Week 222: number analyzed (Participants) | 12
  Week 222 | 85.67 [74.60 to 96.74]
  Week 234: number analyzed (Participants) | 9
  Week 234 | 82.90 [68.16 to 97.63]
  Week 246: number analyzed (Participants) | 7
  Week 246 | 79.83 [61.00 to 98.66]

35. Other Pre Specified Outcome: Change in NEI VFQ-25 Score at Each Study Time Point Relative to Week 8 for Participants Who Had Active Uveitis at Study Entry Over Time
Description: The National Eye Institute (NEI) Visual Functioning Questionnaire (VFQ-25) is an ocular disease-specific survey that measures the influence of visual disability and visual symptoms on generic health domains such as emotional well-being and social functioning, in addition to task-oriented domains related to daily visual functioning.The VFQ-25 consists of a base set of 25 vision-targeted questions plus an additional single-item general health rating question. The overall composite score ranges from 0 to 100, where higher scores or increases in score indicate better vision-related functioning. Baseline was defined as Week 8 for participants with active uveitis.
Time Frame: Weeks 0, 8, 18, 30, 42, 54, 66, 78, 90, 102, 114, 126, 138, 150, 162, 174, 186, 198, 210, 222, 234, and 246
Population: All participants in the ITT analysis set with evaluable data at each timepoint.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 240
score on a scale
  Week 0 | 72.00 [69.52 to 74.48]
  Week 8: number analyzed (Participants) | 226
  Week 8 | 75.77 [73.27 to 78.26]
  Week 18: number analyzed (Participants) | 215
  Week 18 | 78.12 [75.65 to 80.58]
  Week 30: number analyzed (Participants) | 206
  Week 30 | 78.98 [76.46 to 81.50]
  Week 42: number analyzed (Participants) | 197
  Week 42 | 79.77 [77.37 to 82.18]
  Week 54: number analyzed (Participants) | 188
  Week 54 | 80.10 [77.69 to 82.50]
  Week 66: number analyzed (Participants) | 180
  Week 66 | 80.42 [77.87 to 82.97]
  Week 78: number analyzed (Participants) | 169
  Week 78 | 80.98 [78.39 to 83.58]
  Week 90: number analyzed (Participants) | 163
  Week 90 | 81.85 [79.32 to 84.37]
  Week 102: number analyzed (Participants) | 156
  Week 102 | 81.44 [78.74 to 84.14]
  Week 114: number analyzed (Participants) | 146
  Week 114 | 81.76 [78.99 to 84.54]
  Week 126: number analyzed (Participants) | 140
  Week 126 | 81.86 [79.11 to 84.61]
  Week 138: number analyzed (Participants) | 133
  Week 138 | 81.76 [78.94 to 84.59]
  Week 150: number analyzed (Participants) | 123
  Week 150 | 82.41 [79.51 to 85.31]
  Week 162: number analyzed (Participants) | 115
  Week 162 | 81.87 [78.90 to 84.85]
  Week 174: number analyzed (Participants) | 108
  Week 174 | 81.96 [78.78 to 85.14]
  Week 186: number analyzed (Participants) | 97
  Week 186 | 81.27 [78.07 to 84.46]
  Week 198: number analyzed (Participants) | 87
  Week 198 | 82.08 [78.82 to 85.34]
  Week 210: number analyzed (Participants) | 72
  Week 210 | 80.75 [76.99 to 84.51]
  Week 222: number analyzed (Participants) | 59
  Week 222 | 81.65 [77.24 to 86.05]
  Week 234: number analyzed (Participants) | 42
  Week 234 | 81.86 [76.32 to 87.40]
  Week 246: number analyzed (Participants) | 35
  Week 246 | 81.57 [75.44 to 87.70]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until either 70 days after the last dose of study drug or until the first dose of commercially available drug (up to 370 weeks).
Description: TEAEs and SAEs are defined as any AE or SAE with onset or worsening reported by a participant from the time first dose of adalimumab is administered in Study M11-327 until 5 half-lives (70 days) have elapsed following discontinuation of adalimumab or until first dose of commercially available adalimumab post regulatory and/or reimbursement approval for treatment of uveitis in adults in their respective countries. TEAEs were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Adalimumab
All-Cause Mortality (participants affected / at risk) | 4/424
Serious Adverse Events (participants affected / at risk) | 101/424
Other Adverse Events (participants affected / at risk) | 332/424
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab (N=424)
PSEUDOLYMPHOMA (Blood and lymphatic system disorders) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
AORTIC VALVE STENOSIS (Cardiac disorders) | 1 (1)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
BICUSPID AORTIC VALVE (Congenital, familial and genetic disorders) | 1 (1)
BLINDNESS (Eye disorders) | 1 (1)
CATARACT (Eye disorders) | 7 (11)
CILIARY ZONULAR DEHISCENCE (Eye disorders) | 1 (1)
CORNEAL OEDEMA (Eye disorders) | 1 (1)
EYE INFLAMMATION (Eye disorders) | 1 (1)
GLAUCOMA (Eye disorders) | 1 (1)
MACULAR FIBROSIS (Eye disorders) | 1 (1)
OCULAR HYPERTENSION (Eye disorders) | 1 (1)
OPTIC NEUROPATHY (Eye disorders) | 1 (1)
PAPILLOEDEMA (Eye disorders) | 1 (1)
RETINAL DETACHMENT (Eye disorders) | 3 (3)
RETINAL VASCULITIS (Eye disorders) | 1 (1)
UVEITIS (Eye disorders) | 5 (5)
VISUAL ACUITY REDUCED (Eye disorders) | 2 (2)
VITREOUS FLOATERS (Eye disorders) | 1 (1)
VITREOUS HAEMORRHAGE (Eye disorders) | 3 (3)
VITREOUS OPACITIES (Eye disorders) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1)
CROHN'S DISEASE (Gastrointestinal disorders) | 2 (2)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 2 (2)
PANCREATITIS (Gastrointestinal disorders) | 1 (1)
CHEST PAIN (General disorders) | 2 (2)
DEATH (General disorders) | 1 (1)
GENERALISED OEDEMA (General disorders) | 1 (1)
BILIARY COLIC (Hepatobiliary disorders) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 3 (3)
SARCOIDOSIS (Immune system disorders) | 1 (1)
APPENDICITIS (Infections and infestations) | 1 (1)
APPENDICITIS PERFORATED (Infections and infestations) | 1 (1)
ASPERGILLUS INFECTION (Infections and infestations) | 1 (1)
BRAIN ABSCESS (Infections and infestations) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1)
CYTOMEGALOVIRUS CHORIORETINITIS (Infections and infestations) | 1 (2)
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 1 (1)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 2 (3)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 1 (1)
INFECTION (Infections and infestations) | 1 (1)
LATENT TUBERCULOSIS (Infections and infestations) | 1 (1)
MENINGITIS (Infections and infestations) | 1 (1)
OPHTHALMIC HERPES ZOSTER (Infections and infestations) | 1 (1)
PERITONSILLAR ABSCESS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 3 (3)
PYELONEPHRITIS (Infections and infestations) | 2 (2)
PYONEPHROSIS (Infections and infestations) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 1 (1)
SINUSITIS (Infections and infestations) | 2 (2)
SINUSITIS FUNGAL (Infections and infestations) | 1 (1)
SOFT TISSUE INFECTION (Infections and infestations) | 1 (1)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 (1)
TOOTH ABSCESS (Infections and infestations) | 1 (1)
TUBERCULOSIS (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 5 (5)
UROSEPSIS (Infections and infestations) | 1 (1)
COMMINUTED FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
CORNEAL ABRASION (Injury, poisoning and procedural complications) | 1 (1)
ELSCHNIG'S BODIES (Injury, poisoning and procedural complications) | 1 (1)
EPICONDYLITIS (Injury, poisoning and procedural complications) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1)
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 (1)
LACERATION (Injury, poisoning and procedural complications) | 1 (1)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 2 (2)
STRESS FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
CARDIAC MURMUR (Investigations) | 1 (1)
HEPATIC ENZYME INCREASED (Investigations) | 1 (1)
INTRAOCULAR PRESSURE INCREASED (Investigations) | 1 (1)
MYCOBACTERIUM TUBERCULOSIS COMPLEX TEST POSITIVE (Investigations) | 1 (1)
TUBERCULIN TEST POSITIVE (Investigations) | 1 (1)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1)
OBESITY (Metabolism and nutrition disorders) | 3 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
MYOPATHY (Musculoskeletal and connective tissue disorders) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (2)
OSTEOLYSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
PATELLOFEMORAL PAIN SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1)
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
COLORECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
LOBULAR BREAST CARCINOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PANCREATIC CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
RECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
ATAXIA (Nervous system disorders) | 1 (1)
DEMYELINATION (Nervous system disorders) | 1 (1)
ENCEPHALITIS AUTOIMMUNE (Nervous system disorders) | 1 (1)
MULTIPLE SCLEROSIS (Nervous system disorders) | 2 (2)
TENSION HEADACHE (Nervous system disorders) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1)
ECTOPIC PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1 (1)
HYPEREMESIS GRAVIDARUM (Pregnancy, puerperium and perinatal conditions) | 1 (1)
DEVICE DISLOCATION (Product Issues) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1)
BLADDER DIVERTICULUM (Renal and urinary disorders) | 1 (1)
MICTURITION DISORDER (Renal and urinary disorders) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 2 (4)
RENAL COLIC (Renal and urinary disorders) | 1 (1)
URETEROLITHIASIS (Renal and urinary disorders) | 1 (1)
CYSTOCELE (Reproductive system and breast disorders) | 1 (1)
HYDROCELE FEMALE (Reproductive system and breast disorders) | 1 (1)
RECTOCELE (Reproductive system and breast disorders) | 1 (1)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
NASAL POLYPS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1)
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 1 (1)
AORTIC DILATATION (Vascular disorders) | 1 (1)
BEHCET'S SYNDROME (Vascular disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab (N=424)
CATARACT (Eye disorders) | 30 (38)
CYSTOID MACULAR OEDEMA (Eye disorders) | 43 (70)
DRY EYE (Eye disorders) | 30 (33)
EYE PAIN (Eye disorders) | 25 (27)
IRIDOCYCLITIS (Eye disorders) | 22 (29)
MACULAR OEDEMA (Eye disorders) | 24 (31)
UVEITIS (Eye disorders) | 123 (217)
VISUAL ACUITY REDUCED (Eye disorders) | 30 (36)
DIARRHOEA (Gastrointestinal disorders) | 28 (33)
NAUSEA (Gastrointestinal disorders) | 32 (45)
FATIGUE (General disorders) | 36 (42)
PYREXIA (General disorders) | 24 (28)
BRONCHITIS (Infections and infestations) | 38 (50)
INFLUENZA (Infections and infestations) | 36 (44)
NASOPHARYNGITIS (Infections and infestations) | 105 (214)
SINUSITIS (Infections and infestations) | 33 (43)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 43 (65)
URINARY TRACT INFECTION (Infections and infestations) | 47 (66)
INTRAOCULAR PRESSURE INCREASED (Investigations) | 23 (30)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 72 (94)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 26 (30)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 24 (25)
HEADACHE (Nervous system disorders) | 63 (83)
COUGH (Respiratory, thoracic and mediastinal disorders) | 42 (45)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 32 (39)
RASH (Skin and subcutaneous tissue disorders) | 24 (30)
HYPERTENSION (Vascular disorders) | 27 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2015-06-04): https://cdn.clinicaltrials.gov/large-docs/25/NCT01148225/Prot_000.pdf
  • Statistical Analysis Plan (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/25/NCT01148225/SAP_001.pdf